CLINICAL TRIAL: NCT02025179
Title: 12 Month Open-Label Extension Study of the Effect of Teriparatide on Bone in People With Chronic SCI
Brief Title: 12 Month Extension Study of the Effect of Teriparatide on Bone in People With Chronic Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1195
Record Dates: First submitted 2013-12-21; First posted 2013-12-31 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injury; Bone Loss; Osteoporosis
Keywords: Teriparatide; Osteoporosis; Spinal Cord Injury; Bone Diseases; Metabolic Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Nervous System; Wounds and Injuries; Bone Density Conservation Agents; Physiological Effects of Drugs; Pharmacologic Actions; Vibration
MeSH Terms: conditions — Spinal Cord Injuries; Bone Diseases, Metabolic; Osteoporosis; Bone Diseases; Musculoskeletal Diseases; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Wounds and Injuries | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Teriparatide and vibration (Experimental): Experimental: Teriparatide and vibration
  Drug: Teriparatide (Forteo) 20 ug daily Sub-Q over 12 months
  Device: Vibration 10 min/day for 12 months
  Interventions: Drug: Teriparatide; Device: Vibration

INTERVENTIONS:
Drug: Teriparatide — Teriparatide 20 ug daily Sub-Q over 12 months
  Other Names: Forteo
Device: Vibration — Vibration 10 min/day for 12 months
  Other Names: Soloflex Whole Body Vibration platform

SUMMARY:
The purpose of this study is to determine if a second year of exposure to teriparatide in both subjects that received a year of teriparatide or teriparatide-placebo will result in a greater increase in bone mass density (BMD) compared to that seen in a single year's treatment.

This study will also investigate 1) if a second year of teriparatide therapy will increase bone strength in people with chronic spinal cord injury (SCI) who previously received a year of teriparatide or teriparatide-placebo, 2) the number of participants with adverse events from teriparatide, and 3) the effects of teriparatide on serum markers of bone metabolism.

DETAILED DESCRIPTION:
This extension study will only enroll individuals who have completed one year of treatment in the parent protocol "Effect of Teriparatide, Vibration and the Combination on Bone Mass and Bone Architecture in Chronic Spinal Cord Injury (NCT01225055)". This study will allow those individuals who received Teriparatide (20ug/day) and vibration (10 min/day) during the parent study to be treated for a second year and will allow those individuals who received teriparatide-placebo to have the opportunity to have a full year of teriparatide therapy. This study will determine if two years of exposure to teriparatide will result in a greater increase in Bone Mass Density (BMD) than that seen after a single year's treatment. Subjects will be evaluated at 6 and 12 months after initiating treatment with measurement of bone density as well as bone markers of formation and resorption.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in, and completion of one year of treatment, in protocol "Effect of Teriparatide, Vibration and the Combination on Bone Mass and Bone Architecture in Chronic Spinal Cord Injury".
* Adherence rate for teriparatide use of ≥60%.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Individuals who could not tolerate teriparatide treatment.
* Individuals who will not be able to return for all study visits.
* Patients may not be receiving any other investigational agents.
* Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Experimental: Teriparatide and vibration
  Drug: Teriparatide (Forteo) 20 ug daily Sub-Q over 12 months
  Device: Vibration 10 min/day for 12 months
  Completed in previously enrolled study (STU00033380),
  Teriparatide alone with sham vibration
  Teriparatide: 20 ug daily over 12 months
- Vibration: Experimental: Teriparatide and vibration
  Drug: Teriparatide (Forteo) 20 ug daily Sub-Q over 12 months
  Device: Vibration 10 min/day for 12 months
  Completed in previously enrolled study (STU00033380),
  Vibration alone with placebo-teriparatide
  vibration: 10 min/day for 12 months
- Teriparatide and Vibration: Experimental: Teriparatide and vibration
  Drug: Teriparatide (Forteo) 20 ug daily Sub-Q over 12 months
  Device: Vibration 10 min/day for 12 months
  Completed in previously enrolled study (STU00033380),
  Teriparatide with vibration applied in conjunction
  Teriparatide: 20 ug daily over 12 months
  vibration: 10 min/day for 12 months
Period: Overall Study
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Started | 8 | 9 | 8
Completed | 8 | 9 | 7
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration | Total
Number analyzed (Participants) | 8 | 9 | 8 | 25
Age, Continuous [Mean (Full Range); unit: years] | 42.2 [21.1 to 65.3] | 38.0 [22.2 to 62.7] | 41.7 [22.8 to 64.9] | 40.5 [21.1 to 65.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 6 | 7 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 6 | 7 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 5 | 5 | 13
  White | 5 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
American Spinal Injury Association (ASIA) Impairment Scale [Count of Participants; unit: Participants] — ASIA impairment scale describes a person's functional impairment as a result of their spinal cord injury.
  A = Complete. No motor or sensory function in the lowest sacral spine segment (S4-5).
  B = Sensory Incomplete. Sensory function below the neurological level of injury (NLI) and in S4-S5, no motor function below NLI.
  C = Motor Incomplete. Motor function is preserved below NLI and more than half of the key muscle groups below NLI have a muscle grade < 3.
  D = Motor Incomplete. Motor function is preserved below NLI and at least half of the key muscle groups below NLI have a muscle grade 3.
  Participants
    ASIA A (Complete Injury) | 4 | 8 | 7 | 19
    ASIA B (Sensory Incomplete Injury) | 1 | 0 | 1 | 2
    ASIA C (Motor Incomplete Injury) | 3 | 1 | 0 | 4
    ASIA D (Motor Incomplete Injury) | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) of the Total Hip as Assessed by Dual-energy X-ray Absorptiometry (DXA)
Description: The mean percent change in BMD of the total hip after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 7
Percent change | 6.73 [3.37 to 10.1] | -0.34 [-3.50 to 2.82] | 4.24 [0.37 to 8.11]

2. Secondary Outcome: C-terminal Telopeptide
Description: The mean percent change in C-terminal telopeptide from baseline after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 Months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 7
Percent change | -19.8 [-69.0 to 29.5] | -14.8 [-61.2 to 31.6] | -2.12 [-54.8 to 50.5]

3. Secondary Outcome: Bone Mineral Density (BMD) by DXA at the Lumbar Spine
Description: The mean percent change in BMD at the lumbar spine from baseline after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 Months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up. Another subject in "Teriparatide and vibration" spine could not be analyzed due to a baclofen pump.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 6
Percent change | 14.4 [11.0 to 17.8] | 7.05 [3.87 to 10.2] | 8.98 [5.08 to 12.9]

4. Secondary Outcome: Bone Mineral Density (BMD) by DXA at Femoral Neck
Description: The mean percent change in BMD of the femoral neck after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 Months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 7
Percent change | 2.73 [-2.81 to 8.26] | -0.06 [-5.28 to 5.16] | 4.71 [-1.20 to 10.6]

5. Secondary Outcome: Amino-terminal Propeptide of Type 1 Collagen
Description: The mean percent change in Amino-terminal of type 1 collagen from baseline after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 Months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 7
Percent change | 102 [73 to 132] | 104 [76.6 to 132] | 58 [26.6 to 89.5]

6. Secondary Outcome: Bone-specific Alkaline Phosphatase
Description: The mean percent change in Bone-specific alkaline phosphatase from baseline after 24 months of treatment. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section. The "Baseline" refers to the baseline at the parent protocol (NCT01225055). The "24 months" refers to period after the completion of the 12 month parent protocol (NCT01225055) and this 12 month extension study (NCT02025179).
Time Frame: Baseline to 24 Months
Population: One subject in "Teriparatide and vibration" group was lost to follow-up
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 8 | 9 | 7
Percent change | 11.5 [9.04 to 14.0] | 12.6 [10.3 to 14.9] | 10.9 [8.30 to 13.6]

ADVERSE EVENTS:
Time Frame: 12 months
Description: One subject in "Teriparatide and vibration" group was lost to follow-up. Arms/Groups (3) below are divided into the Arms/Groups these subjects were in the parent protocol (NCT01225055) for the 12 month duration of this previous study. These subjects were then enrolled in this 12 month extension study (NCT02025179) and all received Teriparatide and vibration for 12 months as described in the protocol section.
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/9 | 2/7
Other Adverse Events (participants affected / at risk) | 5/8 | 7/9 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=8) | Vibration (N=9) | Teriparatide and Vibration (N=7)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=8) | Vibration (N=9) | Teriparatide and Vibration (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cold/Flu (Infections and infestations) | 2 (3) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cut (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Cut Tip of Left Thumb
Dizziness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Dry scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Lower extremity fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (6)
Pinched nerve (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Pressure sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toe wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No